CLINICAL TRIAL: NCT01719757
Title: A 4-week, Open Label, Multi-center, Prospective, Single-arm, Non-interventional Phase IV Study to Evaluate the Efficacy of Targin for the Treatment of Korean Patients With Cancer Pain Under Conditions of Daily Practice
Brief Title: PROspective Non-interventional Open laBEl Trial for TARGIN in Korean Patients With Cancer Pain
Acronym: PROBE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXN11-KR-404
Record Dates: First submitted 2012-10-08; First posted 2012-11-01 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: Targin, Cancer Pain
MeSH Terms: conditions — Neoplasms; Cancer Pain | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxycodone/naloxone (Experimental): Trade name is Targin. Oxycodone (10mg)/naloxone (5mg) or Oxycodone (20mg)/naloxone (10mg) tablets. Twice daily per oral. Dose adjustment and asymmetric dose are allowed up to 80/40mg per day
  Interventions: Drug: Oxycodone/Naloxone

INTERVENTIONS:
Drug: Oxycodone/Naloxone — Twice daily
  Other Names: Targin

SUMMARY:
The aim of the study is to evaluate the efficacy of TARGIN administration as an analgesic to Korean patients treated with opioid analgesics for moderate-to-severe cancer pain under conditions of daily practice.

DETAILED DESCRIPTION:
An open-label, multi-center, nonrandomized, prospective, non-interventional, observational phase IV trial.

At the first visit, a detailed medical history is taken, including previous analgesics and concomitant treatment. After inclusion, patients enter a 4-week observation period during which they will receive bid of TARGIN 10/5mg and/or 20/10mg. The dose adjustments of TARGIN as well as of analgesic co-medication, rescue-medication and other treatments (e.g. laxatives) can be performed at any time-point during the observation period by the physician in dependence of medical demand. The asymmetric dose is allowed during the observation period by the physician's judgment. (e.g. 10/5 mg in the morning and 20/10 mg in the evening).

Data are gathered using interview-administered questionnaires at baseline (visit 1) and study end (visit 2).

During the observation period, unscheduled visits are allowed after the first visit due to inadequate pain control or occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female cancer patients 20 years of age or older
2. Cancer related pain that requires treatment with continuous around-the-clock strong opioid analgesic
3. Moderate to severe pain intensity (NRS pain score >=4)
4. Opioid naïve patients or patients not treated with strong opioids (Only except occasional PRN) within 13 months or patients who has been on weak opioids
5. Ability to communicate effectively with the study personnel regarding pain intensity, constipation assessment, final assessment of overall efficacy and tolerability
6. Subject who provide signed and dated written voluntary informed consent

Exclusion Criteria:

1. Pregnant or nursing (lactating) women
2. Have previously received treatment with Targin
3. Patient with evidence of significant structural/functional abnormalities of GI tract which is not appropriate for oral medicine administration
4. Any history of hypersensitivity to Oxycodone and Naloxone or any excipients
5. Patients with significant respiratory depression
6. Patients with acute or severe bronchial asthma or hypercarbia
7. Any patient who has or is suspected of having paralytic ileus
8. Severe Chronic obstructive pulmonary disease, pulmonary heart disease
9. Targin product contains lactose. Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not take
10. Patients with moderate and severe hepatic impairment
11. Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), or alkaline phosphatase levels (>2.5 times the upper limit of normal, it is allowed >5 times the upper limit of normal in case of transition in liver) or an abnormal total bilirubin and/or creatinine level(s) (greater than 1.5 times the upper limit of normal)
12. Any situation where opioids are contraindicated
13. With a life expectancy < 1 month
14. Any situation where opioids are contraindicated
15. Mainly pain originated other than cancer or cancer related conditions (eg. Musculoskeletal pain, inflammatory pain, diabetic polyneuropathy)
16. Patients with known or suspected unstable brain metastases or spinal cord compression that may require changes in steroid treatment throughout the duration of the study
17. Patients with uncontrolled seizures
18. Requiring interventional treatment for pain such as neurodestructive procedure or regional infusion
19. With a history of alcohol abuse within 6 months of screening
20. With a history of illicit drug abuse within 6 months of screening
21. Patients with increased intracranial pressure
22. Having used other investigational drugs at the time of enrollment, or within 30 days.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyeonghee Lee, PhD, Principal Investigator — Yeongnam Univ. hospital
Locations (1):
- 13 sites including Yeungnam University Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety set: 359 ITT set: 304
Period: Overall Study
Arm/Group | Oxycodone/Naloxone
Started | 359
Completed | 258
Not Completed | 101
Not completed — Adverse Event | 38
Not completed — Withdrawal by Subject | 15
Not completed — Lost to Follow-up | 20
Not completed — Protocol Violation | 1
Not completed — well controlled pain | 27

BASELINE CHARACTERISTICS:
Population: Safety set
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 359
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 179
  >=65 years | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.73 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 225
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 359

OUTCOME MEASURES:

1. Primary Outcome: Change in Numeric Rating Scales (NRS) Score
Description: Primary objective: Change in numeric rating scales (NRS) such as score for average pain levels over the previous 24 hours, from baseline (visit 1) to study end (visit 2). NRS score was measured from 0 (No pain) to 10(worst pain imaginable).
Time Frame: 4 weeks
Population: Intent to treat analysis set: 304
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 304
units on a scale | -1.89 (2.16)

2. Secondary Outcome: Change of Eastern Cooperative Oncology Group(ECOG) Performance Status
Description: If ECOG P.S score is increased from baseline to visit2, the results mean that QOL was worse.
  ECOG P.S grade: 0=Fully active, able to carry on all pre-disease performance without restriction, 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work,2=Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours,3=Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours,4=Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair,5=Death.
Time Frame: 4weeks
Population: Intent to treat analysis set: 304
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 304
Score | 0.08 (0.52)

3. Secondary Outcome: Change of Constipation Assessment From Baseline to Visit 2(End Visit)
Description: Constipation assessment(5-point scale; 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe, for the patient's judgment of the intensity of symptoms)
Time Frame: 4 weeks
Population: Intent to treat analysis set(Last observational carried forward)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 304
score | -0.03 (0.67)

4. Secondary Outcome: Overall Satisfaction Assessment About Efficacy and Tolerability of Oxycodone/Naloxone by the Investigator and Subject
Description: The overall satisfactions by investigators & subjects were assessed 5 steps such as Very good, Good, Satisfactory, Bad, Very bad.
Time Frame: 4 weeks
Population: Intent to treat analysis set(Last observational carried forward)
Measure: Number; unit: participants
Groups:
- Investigator: For overall satisfaction assessement of oxycodone/naloxone by investigator
- Subject: For overall satisfaction assessement of oxycodone/naloxone by subject
Arm/Group | Investigator | Subject
Number analyzed (Participants) | 304 | 304
participants
  Very good | 24 | 12
  Good | 80 | 78
  Satisfactory | 146 | 156
  Bad | 53 | 55
  Very Bad | 1 | 3

ADVERSE EVENTS:
Time Frame: Safety data were analyzed based on AEs and compliance in the safety set that included subjects who had at least one dose of the study drug and were assessed for safety. Patients were followed safety profile by 4weeks.
Arm/Group | Oxycodone/Naloxone
Serious Adverse Events (participants affected / at risk) | 51/359
Other Adverse Events (participants affected / at risk) | 227/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=359)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Asthenia (General disorders) | 6 (6)
Fatigue (General disorders) | 1 (1)
Disease progression (General disorders) | 4 (4)
Chest discomfort (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=359)
Constipation (Gastrointestinal disorders) | 59 (61)
Nausea (Gastrointestinal disorders) | 48 (52)
Vomiting (Gastrointestinal disorders) | 25 (28)
Diarrhoea (Gastrointestinal disorders) | 22 (29)
Abdominal pain (Gastrointestinal disorders) | 14 (15)
Dyspepsia (Gastrointestinal disorders) | 9 (10)
Stomatitis (Gastrointestinal disorders) | 9 (9)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 24 (33)
Asthenia (General disorders) | 20 (23)
Fatigue (General disorders) | 7 (7)
Chills (General disorders) | 6 (7)
Disease progression (General disorders) | 6 (6)
Chest discomfort (General disorders) | 4 (4)
Oedema (General disorders) | 4 (5)
Pain (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 3 (3)
Catheter site oedema (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 36 (41)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 15 (15)
Headache (Nervous system disorders) | 8 (8)
Hypersomnia (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Speech disorder (Nervous system disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Muscle spasticity (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Oral candidiasis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Furuncle (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 8 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Cold sweat (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 6 (6)
Bladder dilatation (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Flushing (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 4 (4)
Embolism (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (3)
Blood iron decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (7)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No